CLINICAL TRIAL: NCT01695434
Title: A Prospective, Observational, Single-blinded, Longitudinal MRI Study of Effect of Glatiramer Acetate on Iron Deposition in Patients With Relapsing-remitting Multiple Sclerosis Over 24 Months
Brief Title: A Longitudinal Study of Effect of Copaxone in RRMS Over 24 Months
Acronym: GASWI
Status: Completed | Type: Observational
Sponsor: University at Buffalo (Other)
Responsible Party: Principal Investigator, Robert Zivadinov, MD, PhD, Director, Buffalo Neuroimaging Analysis Center, Professor, University at Buffalo
Other Study IDs: GA-SWI 24
Record Dates: First submitted 2012-09-26; First posted 2012-09-28 (Estimated); Last update posted 2013-03-25 (Estimated); Status verified 2013-03

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; MRI; Copaxone; healthy controls; glatiramer acetate
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Copaxone MRI: Patients with relapsing-remitting multiple sclerosis who take Copaxone will have a MRI.
  Interventions: Other: MRI
- Healthy Controls MRI: Subjects who are otherwise healthy, without neurological disorders, will have a MRI.
  Interventions: Other: MRI

INTERVENTIONS:
Other: MRI — All subjects will undergo a MRI.

SUMMARY:
To explore whether treatment with glatiramer acetate (GA) may decrease iron deposition in subcortical deep GM, as detected by SWI-filtered phase imaging, in patients with RRMS over 24 months and compared to a reference population of healthy controls.

DETAILED DESCRIPTION:
This is a prospective, observational, single-blinded, longitudinal, 24-month MRI study of the evolution of iron deposits, as evidenced by SWI-filtered phase imaging, in RRMS patients treated with GA and in healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* MS patients diagnosed with clinically definite MS according to the McDonald criteria (Polman et al., 2005)
* Being on GA monotherapy (20mg/day sc) for at least 24 months prior to the 24-month MRI scan
* Having baseline clinical MRI scan that included SWI-filtered phase imaging in a 12-month window from the start day of the of the GA (MS patients)
* Having baseline clinical MRI scan that included SWI-filtered phase imaging (healthy controls)
* MS patients having a RR disease course (Lublin and Reingold, 1996)
* Age 18-65 (healthy controls will be matched to MS patients for age and sex)
* Signed informed consent at the 24-month follow-up
* Pass MRI health screening
* MS patients passing contrast screening
* MS patients having normal kidney function (creatinine clearance >59)
* None of the exclusion criteria

Exclusion Criteria:

* Patients who had a relapse within 30 days prior to MRI baseline scan date
* Patients who received steroid treatment within 30 days prior to the MRI baseline scan date
* Women who are pregnant, lactating or of childbearing age who do not consent to approved contraceptive use during the study
* MS patients who used other imunomodulatory or immunosuppressant treatment other than GA during the follow-up (e.g., IFN-β, mitoxantrone, cyclophosphamide, cladribine, fludarabine, cyclosporine, total body, azathioprine, methotrexate, IVIG, cellcept, natalizumab, etc.)
* MS patients having abnormal kidney function (creatinine clearance <59)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: MS patients from the Baird MS Center, The Jacobs Neurological Institute, Department of Neurology, State University at Buffalo, NY, USA who are also taking Copaxone as their disease modifying therapy.
  Healthy controls from the general population.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
To explore whether treatment with GA may decrease iron deposition in subcortical deep GM, as detected by SWI-filtered phase imaging, in patients with RRMS over 24 months and compared to a reference population of healthy controls. | 24 months
  MRI collected from RRMS patients who have taken Copaxone for 24 months

SECONDARY OUTCOMES:
To investigate whether treatment with GA may decrease accumulation of iron in lesions, as detected by SWI-filtered phase imaging, in patients with RRMS over 24 months. | 24 months
  Evaluate if Copaxone will decrease iron in lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- Buffalo Neuroimaging Analysis Center, Buffalo, New York, United States